CLINICAL TRIAL: NCT07056868
Title: A Prospective Randomized Controlled Trial Comparing Extraperitoneal Stoma Creation Via the Arcuate Line Approach Versus Conventional Transperitoneal Stoma Formation for the Prevention of Parastomal Hernia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, XIANG ZHANG, Dr., Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: extraperitoneal colostomy
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Parastomal Hernia; Rectal Surgery; Stoma Complications; Extraperitoneal Stoma; Surgical Technique Comparison

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- extraperitoneal colostomy (Experimental): Patients in this group will undergo extraperitoneal stoma creation using the arcuate line approach. This technique involves creating a stoma through the extraperitoneal space by accessing the posterior sheath at or below the arcuate line, thereby avoiding direct peritoneal entry. The goal is to reduce the risk of parastomal hernia by maintaining abdominal wall integrity and preventing intra-abdominal content herniation around the stoma.
  Interventions: Procedure: extraperitoneal colostomy
- transperitoneal colostomy (Active Comparator): Patients in this group will receive a conventional transperitoneal stoma. In this approach, the stoma is brought out through the abdominal wall via a peritoneal opening, which is the standard method used in colorectal surgery. This technique serves as the control for evaluating whether the arcuate line approach offers improved outcomes, particularly in reducing parastomal hernia incidence.
  Interventions: Procedure: transperitoneal colostomy

INTERVENTIONS:
Procedure: extraperitoneal colostomy — Patients in this group will undergo extraperitoneal stoma creation using the arcuate line approach. This technique involves creating a stoma through the extraperitoneal space by accessing the posterior sheath at or below the arcuate line, thereby avoiding direct peritoneal entry. The goal is to reduce the risk of parastomal hernia by maintaining abdominal wall integrity and preventing intra-abdominal content herniation around the stoma.
  Arms: extraperitoneal colostomy
Procedure: transperitoneal colostomy — Patients in this group will receive a conventional transperitoneal stoma. In this approach, the stoma is brought out through the abdominal wall via a peritoneal opening, which is the standard method used in colorectal surgery. This technique serves as the control for evaluating whether the arcuate line approach offers improved outcomes, particularly in reducing parastomal hernia incidence.
  Arms: transperitoneal colostomy

SUMMARY:
This study is a prospective, randomized controlled trial designed to compare two surgical techniques for stoma creation in patients undergoing colorectal surgery. The trial evaluates whether an extraperitoneal stoma created via the arcuate line approach can reduce the risk of developing parastomal hernia compared to the conventional transperitoneal stoma formation. Parastomal hernia is a common complication after stoma surgery, often requiring additional treatment or surgery. By testing a novel surgical route that avoids entering the abdominal cavity, this study aims to improve postoperative outcomes and quality of life for patients requiring a permanent stoma.

DETAILED DESCRIPTION:
Parastomal hernia (PSH) is one of the most common long-term complications following stoma creation, with incidence rates reported as high as 30-50%. Conventional stoma formation typically uses a transperitoneal route, which may leave potential gaps in the abdominal wall through which herniation can occur.

Recent anatomical and surgical advances have proposed the arcuate line approach for extraperitoneal stoma creation, allowing the stoma to be tunneled outside the peritoneal cavity while preserving abdominal wall integrity. However, robust prospective evidence supporting its clinical benefits remains limited.

This randomized controlled trial will compare the arcuate line extraperitoneal approach with the traditional transperitoneal method, focusing on the incidence of parastomal hernia as the primary outcome. Secondary outcomes include postoperative complications, operative time, stoma function, and quality of life.

The results may provide high-level evidence to guide best practices in stoma surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Scheduled for laparoscopic abdominoperineal resection

Written informed consent

Exclusion Criteria:

* Previous abdominal wall hernia

Emergency surgery

Severe comorbidities prohibiting safe surgery

Prior lower abdominal surgery affecting stoma site

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Parastomal Hernia | 36 months postoperatively
  The occurrence of parastomal hernia will be assessed at 36 months after surgery through both clinical examination and abdominal CT imaging. Parastomal hernia will be defined based on radiological criteria (e.g., herniation of abdominal contents adjacent to the stoma) and/or physical examination findings (bulging or protrusion around the stoma site). The primary endpoint is the proportion of patients in each group who develop parastomal hernia within the follow-up period.

IPD SHARING:
Plan to Share IPD: No